CLINICAL TRIAL: NCT05147207
Title: Supercapsular Percutaneously-Assisted Total Hip (SuperPATH®) Versus Conventional Posterior Approach for Total Hip Arthroplasty: A Prospective Randomized Controlled Study
Brief Title: SuperPath Versus Posterior Approach for THA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Gavin Wood, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SURG-387-17
Record Dates: First submitted 2021-10-20; First posted 2021-12-07 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Surgical Approach; Hip Arthropathy

STUDY DESIGN:
Intervention Model Description: superpath approach versus posterior approach
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Superpath (Experimental): This is a minimally invasive surgical approach.
  Interventions: Procedure: Superpath Approach
- Posterior Approach (No Intervention): This is the traditional THA surgical approach used.

INTERVENTIONS:
Procedure: Superpath Approach — This is a minimally invasive surgical approach for THA.
  Arms: Superpath

SUMMARY:
The SuperPATH approach is a minimally invasive approach for total hip arthroplasty. This project randomized patients to the SuperPath versus posterior approach. Outcomes examined included functional, VAS pain, narcotic utilization, perioperative outcomes, and radiographic component positions. Participants were followed for 2 years. The aim was to examine if the SuperPATH approach provided significant advantages over the posterior approach on functional testing or return to work for patients.

DETAILED DESCRIPTION:
Background: The Supercapsular Percutaneously-Assisted Total Hip (SuperPATH) approach is a minimally invasive approach for total hip arthroplasty. It has been reported to show earlier mobilization, better gait kinematics, and short hospital length of stay. Our primary objective was to compare functional tests of timed up and go and timed stair climb preoperatively, at discharge, 2 weeks, and 6 weeks postoperatively. Secondary objectives included the return to function in weeks, Oxford hip scores, visual analog scale, narcotic utilization, perioperative outcomes, and radiographic component positions.

Methods: Forty-six patients were randomized into two groups on the surgery day: the SuperPATH group (25 patients) and the Posterior group (20 patients). Outcomes examined included functional, VAS pain, narcotic utilization, perioperative outcomes, and radiographic component positions.

ELIGIBILITY:
Inclusion Criteria:

* Non-inflammatory degenerative joint disease including osteoarthritis, traumatic arthritis, or avascular necrosis;
* Inflammatory degenerative joint disease including rheumatoid arthritis;
* Correction of functional deformity.
* Subject is skeletally mature (21 years of age or older);
* Subject is a candidate to be implanted with the specified combination of components;
* Subject is willing and able to complete required study visits and assessments;
* Subject plans to be available through the follow-up visits;
* Subject is willing to sign the approved informed consent document.
* Subjects with a previous THA in the contralateral hip are eligible for enrollment provided it has been at least 1 year since the contralateral THA and the contralateral THA is asymptomatic and not pending revision. Simultaneous bilateral THA subjects will not be permitted to enroll.

Exclusion Criteria:

* Subject has overt infection or distant foci of infections;
* Subject has rapid disease progression as manifested by joint destruction or bone absorption apparent on roentgenogram;
* Subject with inadequate neuromuscular status (e.g. prior paralysis, fusion and/or inadequate abductor strength), poor bone stock, poor skin coverage around the joint which would make the procedure unjustifiable;
* Subject has a neuropathic joints;
* Subject has hepatitis or HIV infection;
* Subject has a neurological or musculoskeletal disease that may adversely affect gait or weight-bearing;
* Subject is currently enrolled in another clinical investigation that could affect the endpoints of this study;
* Subject is unwilling or unable to sign the informed consent document;
* Subject has documented substance abuse issues;
* Subject has a body mass index (BMI) of greater than 40;

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Functional Outcomes TUG | 6 weeks
  Timed up and go test
Functional Outcomes TSC | 6 weeks
  Timed stair climb

SECONDARY OUTCOMES:
Subjective Measure | 3 months
  Oxford Hip Score - score from 0 (severe hip arthritis) to 48 (satisfactory joint function)
Pain Score | 1 month
  Visual Analog Scale - score from 0 (no pain) to 10 (worst pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khoja YT, Habis AA, Wood GCA. The Supercapsular Percutaneously Assisted Total Hip Approach Does Not Provide Any Clinical Advantage Over the Conventional Posterior Approach for THA in a Randomized Clinical Trial. Clin Orthop Relat Res. 2023 Jun 1;481(6):1116-1125. doi: 10.1097/CORR.0000000000002449. Epub 2022 Nov 8. PMID 36350098